CLINICAL TRIAL: NCT04495725
Title: Do Discounted Vouchers for Medical Cannabis Reduce Opioid Use in Adults With Pain: A Randomized Controlled Trial (The ReLeaf-V Study)
Brief Title: Do Discounted Vouchers for Medical Cannabis Reduce Opioid Use in Adults With Pain
Acronym: ReLeaf-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vireo Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ReLeaf-V
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use; Marijuana; Chronic Pain
Keywords: opioid; marijuana; cannabis; pain
MeSH Terms: conditions — Marijuana Abuse; Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Voucher for a Discounted Placebo Product (Placebo Comparator): Voucher for a Discounted Placebo Soft-Gel Capsule Product
  Interventions: Other: Discounted Vouchers for Medical Cannabis Soft-Gel Capsule Products
- Voucher for a Discounted High THC:Low CBD Product (Experimental): Voucher for a Discounted 4.3mg THC/0.7mg CBD Soft-Gel Capsule Product
  Interventions: Other: Discounted Vouchers for Medical Cannabis Soft-Gel Capsule Products
- Voucher for a Discounted Equal THC:CBD Product (Experimental): Voucher for a Discounted 2.5mg THC/2.5mg CBD Soft-Gel Capsule Product
  Interventions: Other: Discounted Vouchers for Medical Cannabis Soft-Gel Capsule Products
- Voucher for a Discounted Low THC:High CBD Product (Experimental): Voucher for a Discounted 0.2mg THC/4.8mg CBD Soft-Gel Capsule Product
  Interventions: Other: Discounted Vouchers for Medical Cannabis Soft-Gel Capsule Products

INTERVENTIONS:
Other: Discounted Vouchers for Medical Cannabis Soft-Gel Capsule Products — We will randomize participants to one of the following four conditions for discounted vouchers: 1) a discounted voucher for a placebo soft-gel capsule product, 2) a discounted voucher for a high THC:low CBD soft-gel capsule product, 3) a discounted voucher for an equal THC:CBD soft-gel capsule product, or 4) a discounted voucher for a low THC:high CBD soft-gel capsule product. We will stratify randomization by history of cannabis use (no use in the past year, used in the past year and not near-daily or daily (used in the past year and <20 days out of the last 30 days), near-daily or daily (>= 20 days out of the last 30 days) baseline opioid analgesic prescription (chronic opioid treatment vs. not chronic opioid use), and primary pain condition (neuropathy, not neuropathy). Chronic opioid treatment is defined as prescribed opioids ≥90 non-overlapping days in the past 182 days. Randomization will occur in blocks to ensure equal randomization over time.

SUMMARY:
This study will examine how discounted vouchers for medical cannabis use affects opioid analgesic use in adults with chronic pain. Our study findings will have critically important implications to shape clinical care and medical cannabis policies.

DETAILED DESCRIPTION:
This study will examine how discounted vouchers for medical cannabis use affects opioid analgesic use in adults with chronic pain. ReLeaf-V is a 4-arm blinded randomized controlled trial (RCT) of 352 adults with (a) severe or chronic neuropathic or joint pain, (b) opioid analgesic use, and (c) active certification for medical cannabis. We will randomize participants to a discounted voucher for: 1) a placebo soft-gel capsule product, 2) high THC:low CBD soft-gel capsule product (4.3mg THC/0.7mg CBD), 3) equal THC:CBD soft-gel capsule product (2.5mg THC/2.5mg CBD), or 4) low THC:high CBD soft-gel capsule product (0.2mg THC/4.8mg CBD). Over 14 weeks, participants will have 5 research visits in which data will be collected from questionnaires, and medical and Prescription Monitoring Program (PMP) records. The primary independent variable will be randomization arm, and the primary outcome will be cumulative opioid analgesic dose.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. English or Spanish fluency
3. active certification for medical cannabis
4. intends to have a soft-gel capsule product dispensed at Vireo Health
5. medical cannabis qualifying conditions or complications of (a) chronic pain, or (b) pain that degrades health and functional capability as an alternative to opioid use or substance use disorder or (c) severe or chronic pain
6. joint or neuropathic pain
7. current severe pain
8. dispensed opioids analgesics within the last 60 days

To maintain the integrity of the study, we do not disclose all inclusion criteria to potential participants.

Exclusion Criteria:

1. inability to provide informed consent
2. inability to complete study visits over 14 weeks
3. terminal illness
4. current or prior psychotic disorder
5. current or prior buprenorphine or methadone treatment for opioid use disorder
6. NYS medical marijuana prescriber does not approve changes to product and dosing recommendations listed on the participant's certification form
7. Allergy to tapioca or coconut
8. currently pregnant, planning to become pregnant within the next 3 months, or breastfeeding
9. a condition that is considered by a pharmacist or medical provider to be a clinical contraindication to medical cannabis use (e.g. unstable cardiac arrhythmia or specific drug-drug interaction)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Opioid analgesic use | Opioid analgesic use will be weekly cumulative dose of opioid analgesics over 14 weeks.
  The primary outcome will be cumulative opioid analgesic dose.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dahmer, MD, Principal Investigator — Vireo Health of New York; Giovanna DiFrancesca, Study Director — Albert Einstein College of Medicine
Locations (1):
- Vireo Health of New York, Queens, New York, United States